CLINICAL TRIAL: NCT00658775
Title: A Randomized, Double-Blind, Parallel Study of Rabeprazole Extended-Release 50 mg Versus Esomeprazole 40 mg for Healing and Symptomatic Relief of Moderate to Severe Erosive Gastroesophageal Reflux Disease (GERD)
Brief Title: Rabeprazole Extended-Release, 50 mg, Versus Esomeprazole, 40 mg, for Healing and Symptomatic Relief of Moderate to Severe Erosive Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3810-G000-302; 2007-006046-17 (EudraCT Number)
Record Dates: First submitted 2008-04-09; First posted 2008-04-15 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: GERD; erosive GERD; erosive esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Rabeprazole sodium
- 2 (Active Comparator)
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Rabeprazole sodium — Rabeprazole ER 50 mg capsule, once daily for 4-8 weeks.
  Other Names: Aciphex
  Arms: 1
Drug: Esomeprazole — Esomeprazole 40 mg capsule, once daily for 4-8 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the efficacy (ie, healing and symptom relief) and safety of Rabeprazole Extended-Release (RAB ER) 50 mg versus Esomeprazole (ESO) 40 mg for the treatment of moderate to severe erosive Gastroesophageal Reflux Disease (eGERD).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, double-dummy, parallel-group study. Subjects who meet all the inclusion/exclusion criteria will be randomly assigned to 1 of 2 treatment groups, Rabeprazole Extended-Release (RAB ER) 50 mg or Esomeprazole (ESO) 40 mg for the treatment of moderate to severe erosive Gastroesophageal Reflux Disease (eGERD).

ELIGIBILITY:
KEY INCLUSION CRITERIA:

1. Male or female, ages 18 to 75 years.
2. History of GERD symptoms for at least 3 months immediately before screening.
3. Heartburn for at least 2 days a week for at least 1 month before screening.
4. Esophageal erosions of LA Grades C or D based on EGD taken within 14 days prior to enrollment.
5. Subjects who are H. pylori negative based on a screening test.
6. Females should be either of non-childbearing potential or of childbearing potential. Females of childbearing potential must have negative pregnancy tests prior to randomization. Female subjects of childbearing potential must agree to use medically acceptable methods of contraception.
7. Subjects must be able to read, write, and understand the language of the symptom diary.

KEY EXCLUSION CRITERIA:

1. Current or a history of esophageal motility disorders.
2. Current or a history of Barrett's esophagus.
3. Current esophageal strictures or esophagitis (known or suspected to be due to etiology other than GERD such as infection or medications).
4. Current or a history of Zollinger-Ellison syndrome and other acid hypersecretory conditions, or current gastric or duodenal ulcer.
5. Current or a history of cancer, with the exception of fully excised skin basal cell carcinoma.
6. Inflammatory bowel disease.
7. Unstable diabetes mellitus.
8. History of esophageal, gastric and duodenal surgery except simple suturing of an ulcer.
9. Subjects who require daily use of nonsteroidal anti-inflammatory drugs (NSAIDs), oral steroids (>= 20 mg/day prednisone or equivalent), or aspirin (> 325 mg/day).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1069 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yufang Lu, Study Director — Eisai Inc.
Locations (68):
- Moline, Illinois, United States
- Argentina (5):
  - La Plata, Argentina
  - Buenos Aires, BUE
  - Ciudad Autonoma de Bs. As., CBA
  - Rosario, SFE
  - San Miguel de Tucumán, TUC
- Australia (7):
  - Penrith, New South Wales
  - Caboolture, Queensland
  - Adelaide, South Australia
  - Woodville, South Australia
  - Launceston, Tasmania
  - Ballarat, Victoria
  - Fitzroy, Victoria
- Bulgaria (4):
  - Haskovo, Bulgaria
  - Plovdiv, Bulgaria
  - Rousse, Bulgaria
  - Sofia, Bulgaria
- Canada (8):
  - Barrie, Ontario
  - Chatham, Ontario
  - Hamilton, Ontario
  - Richmond Hill, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Sherbrooke, Quebec
  - Saskatoon, Saskatchewan
- Chile (3):
  - Providencia, Chile
  - Santiago, Chile
  - Temuco, Chile
- Croatia (3):
  - Osijek, Croatia
  - Split, Croatia
  - Zagreb, Croatia
- Tallinn, Estonia, Estonia
- France (3):
  - Saint-Quentin, France
  - Lyon, Lyonnais
  - Marseille, Provence-Alpes-Côte d'Azur Region
- Germany (8):
  - Freising, Bavaria
  - Potsdam, BR
  - Herne, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Ludwigshafen am Rhein, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Wolmirstedt, Saxony-Anhalt
- Hungary (10):
  - Balatonfüred, Hungary
  - Budapest, Hungary
  - Debrecen, Hungary
  - Eger, Hungary
  - Győr, Hungary
  - Gyula, Hungary
  - Kaposvár, Hungary
  - Pécs, Hungary
  - Siófok, Hungary
  - Szekszárd, Hungary
- India (10):
  - Hyderabad, Andhra Pradesh
  - Secunderabad, Andhra Pradesh
  - Visakhapatnam, Andhra Pradesh
  - Bangalore, Karnataka
  - Mangalore, Karnataka
  - Kochi, Kerala
  - New Delhi, National Capital Territory of Delhi
  - Ludhiana, Punjab
  - Chennai, Tamil Nadu
  - Madurai, Tamil Nadu
- Latvia (3):
  - Balvi, Latvia
  - Daugavpils, Latvia
  - Riga, Latvia
- Lithuania (2):
  - Šiauliai, Lithuania
  - Vilnius, Lithuania

REFERENCES:
- [Derived] Laine L, Katz PO, Johnson DA, Ibegbu I, Goldstein MJ, Chou C, Rossiter G, Lu Y. Randomised clinical trial: a novel rabeprazole extended release 50 mg formulation vs. esomeprazole 40 mg in healing of moderate-to-severe erosive oesophagitis - the results of two double-blind studies. Aliment Pharmacol Ther. 2011 Jan;33(2):203-12. doi: 10.1111/j.1365-2036.2010.04516.x. Epub 2010 Nov 30. PMID 21114792

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 1069 participants who were randomized, 1065 participants received study treatment.
Groups:
- ESO 40mg: Esomeprazole (ESO) 40mg capsule concurrently with placebo (identical in appearance to the RAB Extended Release (ER) 50mg capsule), once daily for 4 to 8 weeks.
- RAB ER 50mg: Rabeprazole (RAB) Extended Release (ER) 50mg capsule concurrently with placebo (identical in appearance to the ESO 40mg capsule), once daily for 4 to 8 weeks.
Period: Overall Study
Arm/Group | ESO 40mg | RAB ER 50mg
Started | 537 (Treated) | 528 (Treated)
Completed | 495 | 485
Not Completed | 42 | 43
Not completed — Adverse Event | 4 | 6
Not completed — Lost to Follow-up | 17 | 18
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Withdrawal of consent | 8 | 7
Not completed — Other | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESO 40mg | RAB ER 50mg | Total
Number analyzed (Participants) | 537 | 528 | 1065
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.1 (13.38) | 51 (12.79) | 50 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 179 | 374
  Male | 342 | 349 | 691

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Who Achieved Diary-recorded Sustained Resolution of Heartburn by Week 4
Description: During the first 4 weeks of the Double-blind Phase, participants were to record heartburn in a daily diary. Participant daily symptoms for the assessment of heartburn was based on a commonly used 4-point Likert scale of none, mild, moderate and severe. A participant was considered achieving sustained resolution of heartburn if the participant had maintained at least 7 consecutive heartburn-free days.
Time Frame: Week 4
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | ESO 40mg | RAB ER 50mg
Number analyzed (Participants) | 537 | 528
Percentage of Participants
  Yes | 52.5 | 53.2
  No | 40 | 39.6
  Missing | 7.4 | 7.2

2. Primary Outcome: Percentage of Participants With Erosive Gastroesophageal Reflux Disease (eGERD) Who Achieved Endoscopically-confirmed Healing by 8 Weeks
Description: Healing at week 4 or 8 were based on improvement of eGERD of the Los Angeles (LA) classification of esophagitis Grade C or D from Baseline. Classifications include:
  Not Present: No breaks (erosions) in the esophageal mucosa (however, edema, erythema, or friability may be present) Grade A: One or more mucosal breaks not more than 5mm in maximum length. Grade B: One or more mucosal breaks more than 5mm in maximum length, but not continuous between the tops of 2 mucosal folds.
  Grade C: Mucosal breaks continuous between the tops of 2 or more mucosal folds, but involving less than 75% of the esophageal circumference.
  Grade D: Mucosal breaks involving at least 75% of the esophageal circumference.
Time Frame: Baseline and Week 8
Population: ITT Population - all randomized subjects who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | ESO 40mg | RAB ER 50mg
Number analyzed (Participants) | 537 | 528
Percentage of Participants
  Yes | 78.4 | 77.5
  No | 16.6 | 18.4
  Missing | 5 | 4.2

3. Primary Outcome: Percentage of Participants With eGERD Who Achieved Endoscopically-confirmed Healing by 4 Weeks
Description: Healing at week 4 or 8 were based on improvement of eGERD of the LA classification of esophagitis Grade C or D from Baseline. Classifications include:
  Not Present: No breaks (erosions) in the esophageal mucosa (however, edema, erythema, or friability may be present) Grade A: One or more mucosal breaks not more than 5mm in maximum length. Grade B: One or more mucosal breaks more than 5mm in maximum length, but not continuous between the tops of 2 mucosal folds.
  Grade C: Mucosal breaks continuous between the tops of 2 or more mucosal folds, but involving less than 75% of the esophageal circumference.
  Grade D: Mucosal breaks involving at least 75% of the esophageal circumference.
Time Frame: Baseline and Week 4
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | ESO 40mg | RAB ER 50mg
Number analyzed (Participants) | 537 | 528
Percentage of Participants
  Yes | 50.7 | 50.9
  No | 46.4 | 47
  Missing | 3 | 2.1

ADVERSE EVENTS:
Time Frame: For each participant, from the time of administration of the first dose of study drug up to 30 days after the administration of the last dose of study drug or up to resolution of adverse event or up to approximately 10 weeks.
Description: Data are presented as number of participants with treatment emergent adverse events (serious and nonserious). The analysis was performed using Safety Analysis Set (SAS) defined as all subjects who received at least 1 dose of study drug and had a postbaseline safety assessment.
Arm/Group | ESO 40mg | RAB ER 50mg
Serious Adverse Events (participants affected / at risk) | 3/532 | 3/526
Other Adverse Events (participants affected / at risk) | 0/532 | 0/526
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ESO 40mg (N=532) | RAB ER 50mg (N=526)
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No